CLINICAL TRIAL: NCT04057131
Title: FIRAZYR General Drug Use-Results Survey (Japan)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP667-401
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firazyr: Participants with Hereditary angioedema (HAE) receiving treatment with Icatibant acetate (Firazyr) as prescribed by their physician following locally approved prescribing information.
  Interventions: Drug: Firazyr

INTERVENTIONS:
Drug: Firazyr — Participants with Hereditary angioedema (HAE) receiving treatment with Icatibant acetate (Firazyr) as prescribed by their physician following locally approved prescribing information.
  Other Names: Icatibant acetate

SUMMARY:
The objectives of this survey are to collect data to report the safety and efficacy of Firazyr (Icatibant acetate) in the post-marketing phase in participants diagnosed with Hereditary Angioedema (HAE).

ELIGIBILITY:
Inclusion Criteria:

* Hereditary angioedema (HAE) participants in Japan who receive FIRAZYR for first time in the real world clinical setting.

Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hereditary angioedema (HAE) patients in Japan who receive FIRAZYR for first time in the real world clinical setting are eligible for enrollment in this survey.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (18):
- Japan (18):
  - Nagoya-city, Nagoya, Aichi-ken
  - Toyohashi-city, Toyohashi, Aichi-ken
  - Maebashi-city, Maebashi, Gunma
  - Asahikawa-city, Asahikawa, Hokkaido
  - Fukagawa-city, Fukagawa, Hokkaido
  - Rumoi-city, Rumoi, Hokkaido
  - Sapporo-city, Sapporo, Hokkaido
  - Kasama-city, Kasama, Ibaraki
  - Maizuru-city, Maizuru, Kyoto
  - Kishiwada-city, Kishiwada, Osaka
  - Takatsuki-city, Takatsuki, Osaka
  - Kawagoe-city, Kawagoe, Saitama
  - Soka-city, Sōka, Saitama
  - Numazu-city, Numazu, Shizuoka
  - Shimada-city, Shimada, Shizuoka
  - Yaezu-city, Yaezu, Shizuoka
  - Tachikawa-city, Tachikawa, Tokyo
  - Niigata-city, Niigata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47b02

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 93 investigative sites in Japan, from 20 Nov 2018 to 29 Jul 2024.
Pre-assignment Details: Participants with Hereditary Angioedema (HAE) received Icatibant acetate subcutaneous infusion as part of a routine medical care.
Groups:
- Icatibant Acetate Subcutaneous Infusion: Participants with Hereditary Angioedema (HAE) received Icatibant acetate subcutaneous infusion as part of a routine medical care.
Period: Overall Study
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Started | 179
Completed | 155
Not Completed | 24
Not completed — Protocol Violation | 24

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number analyzed is the number of participants with data available for analysis.
  years
    number analyzed (Participants) | 151
    (all) | 41.6 (15.3)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Unknown: Data could not be collected.
  Participants
    Female | 116
    Male | 38
    Unknown | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Baseline up to end of the study (up to approximately 68 months)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 155
Participants | 22

2. Primary Outcome: Number of Participants With Adverse Drug Reaction
Description: An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. Adverse drug reaction refers to AE related to administered drug.
Time Frame: Baseline up to end of the study (up to approximately 68 months)
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 155
Participants | 19

3. Primary Outcome: Time to Treatment for Attack
Description: Time to treatment for attack defined as the time between the onset of the attack and the first injection of treatment. Time to treatment for attack was assessed and reported.
Time Frame: Up to 3 months
Population: Efficacy analysis set: all participants who received at least one dose of protocol treatment without major protocol deviation.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 100
minutes | 120.0 [30.0 to 360.0]

4. Primary Outcome: Time to First Symptom Relief
Description: Time to first symptom relief defined as the time between the first injection of treatment and first symptom relief. Time to first symptom relief was assessed and reported.
Time Frame: Up to 3 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 100
minutes | 60.0 [30.0 to 450.0]

5. Primary Outcome: Time to Complete Resolution of Attack
Description: Time to complete resolution of attack defined as the time between the first injection of treatment and the complete resolution of all symptoms. Time to complete resolution of attack was assessed and reported.
Time Frame: Up to 3 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 100
minutes | 780.0 [210.0 to 1800.0]

6. Primary Outcome: Total Duration of Attack
Description: Total duration of attack defined as the time between the onset of the attack and the complete resolution of all symptoms. Total duration of attack was assessed and reported.
Time Frame: Up to 3 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Icatibant Acetate Subcutaneous Infusion
Number analyzed (Participants) | 100
minutes | 1425.0 [420.0 to 2880.0]

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (up to approximately 68 months)
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Icatibant Acetate Subcutaneous Infusion
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 1/155
Other Adverse Events (participants affected / at risk) | 7/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Icatibant Acetate Subcutaneous Infusion (N=155)
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Icatibant Acetate Subcutaneous Infusion (N=155)
Injection site pain (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04057131/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT04057131/SAP_001.pdf